CLINICAL TRIAL: NCT02377492
Title: Paracervical Vasopressin Injection Compared With Intramyometrial Vasopressin in Abdominal Myomectomy: A Randomized Controlled Trial
Brief Title: Paracervical Vasopressin Injection Compared With Intramyometrial Vasopressin in Abdominal Myomectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 043231
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracervical & Intramyometrial (Experimental): Vasopressin will be placed paracervically (8mL, 4 units) and intramyometrial (8mL, 4 units)
  Interventions: Drug: Vasopressins
- Intramyometrial (Active Comparator): Vasopressin will be placed intramyometrial (16mL, 8 units)
  Interventions: Drug: Vasopressins

INTERVENTIONS:
Drug: Vasopressins — Either paracervical and intramyometrial or intramyometrial alone at time of abdominal myomectomy.
  Other Names: vasopressin

SUMMARY:
The goal of the investigators study is to evaluate the effectiveness of paracervical injection of vasopressin at the time of abdominal myomectomy to decrease blood loss. The investigators will continue to use intramyometrial vasopressin as this has previously been shown to be effective. The study will not exceed the safely documented dose of vasopressin.

DETAILED DESCRIPTION:
After the initial physician consultation and investigations have been completed, the treatment options will be reviewed with the patient. If the patient chooses to proceed with an abdominal myomectomy, then she will be offered participation in the study.

If she chooses to participate, the patient will undergo routine pre-operative assessments including either transvaginal ultrasound or pelvic MRI. The pre-operative hemoglobin level will be measured within at least 2 weeks of the operative procedure.

Randomization to either the vasopressin group or the placebo group will be carried out in the operating room by assigning each recruited patient a consecutively numbered, sealed opaque envelope, which will contain the designated treatment as determined by a computer-generated series of random numbers. The randomization will be performed by an independent member of the division that is not involved in the study.

At the time of induction of anesthesia, a sealed envelope will be opened by the research fellow. At the time of induction of anesthesia, the sealed envelope will be opened to reveal the randomization to only the research fellow. The attending physician will remain blinded. The research fellow will prepare either the placebo solution or the vasopressin and will be responsible for performing the paracervical injection. The attending physician will be responsible for recording the surgeon rate of bleeding, the total ebl, and the total operating time.

In the both groups, one vial (20 units) of vasopressin will be diluted to 40mL with normal saline solution. Not more than 16mL (8units) of vasopressin will be used. This dose was chosen as there is no standard vasopressin dose routinely used. The dose is well below the maximum amount of vasopressin used, and at a level that few complications have been seen in the past.

Given it is standard practice for all patients to receive intramyometrial vasopressin injections, both groups will have the medication ordered and prepared. In the patients randomized to paracervical vasopressin, 8mL (4mL per side of the cervix) will be injected using a 22F spinal needle. An additional 8mL (4 units) will be injected in intramyometrial as this is standard of care in our practice. In the patients randomized to no paracervical vasopressin, 16mL (8 units) will then be used to inject vasopressin intramyometrial prior to the myomectomy. This will help determine if the routine of delivery of vasopressin will aid in decreased blood loss.

The operative case will otherwise proceed in the standard fashion. The total ebl, total operative time, and myomectomy operative time will all be recorded. The myomectomy operative time will be recorded from the time of the first incision on the uterus, to complete closure of any uterine defects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* All women who are candidates for abdominal myomectomy and are willing to accept randomization

Exclusion Criteria:

* Patients unable to consent for the study
* Suspected malignancy
* History of adverse reaction or allergy to vasopressin
* Active cardiovascular or pulmonary disease that would indicate a contraindication to use of vasopressin

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
1. Estimating blood loss at the end of myomectomy (calculated as [total suction canister volume] +[laparotomy pads] - [volume of irritation used] - [volume of vasopressin used]) | 1 day

SECONDARY OUTCOMES:
Change in Hgb and Hct post-operatively from pre-operative level | 1- 2 days
Peri-operative complications | 2 days
Total operation time (time from incision to end of surgery) | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Hospitals Fertility Center, Beachwood, Ohio
  - University Hospitals, Cleveland, Ohio